CLINICAL TRIAL: NCT00379704
Title: TIFACT Study - Tissue Factor Expression by Adipose Tissue in Extremely Obese Subjects. Relationship With Circulating Tissue Factor and Coagulation Activation Markers
Brief Title: TIFACT Study - Tissue Factor Expression by Adipose Tissue in Extremely Obese Subjects.
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P060307
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2007-03

CONDITIONS: Obesity
Keywords: Tissue factor; Obesity; Adipose tissue; Microparticles
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — samples of plasma and serum and greasy fragments
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Tissue factor is the main activator of coagulation cascades. Excessive tissue factor expression is made responsible of thrombosis in a number of clinical situations including thrombosis in contact with atherosclerotic plaques. Recent work showed that tissue factor gene expression in adipose tissue was significantly increased in obese versus lean mice.

The main objective of this study is to show that tissue factor expression is increased in human adipose tissue obtained from obese subjects and to identify its main tissular origin by comparing abdominal and subcutaneous adipose tissue.

The secondary objectives are to identify the cell origin of tissue factor (adipocytes versus stromal cells) and to analyze the relation ship between blood tissue factor and (i) tissue factor expressed by adipose tissue, (ii) the amount of subcutaneous and profound adipose tissue, and (iii) coagulation activation markers.

DETAILED DESCRIPTION:
Tissue factor is the main activator of coagulation cascades. Excessive tissue factor expression is made responsible of thrombosis in a number of clinical situations including thrombosis in contact with atherosclerotic plaques. Recent work showed that tissue factor gene expression in adipose tissue was significantly increased in obese versus lean mice.

The main objective of this study is to show that tissue factor expression is increased in human adipose tissue obtained from obese subjects and to identify its main tissular origin by comparing abdominal and subcutaneous adipose tissue.

The secondary objectives are to identify the cell origin of tissue factor (adipocytes versus stromal cells) and to analyze the relation ship between blood tissue factor and (i) tissue factor expressed by adipose tissue,

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35
* Stable obesity
* Abdominal or pelvic surgery
* Agree to participate to the study

Exclusion Criteria:

* malignancy,
* infectious or inflammatory disease, notably HIV infection
* pregnancy
* history of ischemic cardio or neurovascular event, lower limb arteritis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inclusion Criteria:
  * BMI > 35
  * Stable obesity
  * Abdominal or pelvic surgery
  * Agree to participate to the study
  Exclusion Criteria:
  * malignancy,
  * infectious or inflammatory disease, notably HIV infection
  * pregnancy
  * history of ischemic cardio or neurovascular event, lower limb arteritis
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2006-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain STEPANIAN, MD PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- CHU Louis Mourier, Colombes, France

REFERENCES:
- [Background] Samad F, Pandey M, Loskutoff DJ. Regulation of tissue factor gene expression in obesity. Blood. 2001 Dec 1;98(12):3353-8. doi: 10.1182/blood.v98.12.3353. PMID 11719374